CLINICAL TRIAL: NCT00463385
Title: A Phase 2, Prospective, Randomized, Multicenter, Double-blind, Active-control, Parallel-group Study to Determine the Safety of and to Select a Treatment Regimen of CC-4047 (Pomalidomide) Either as Single-agent or in Combination With Prednisone to Study Further in Subjects With Myelofibrosis With Myeloid Metaplasia
Brief Title: A Phase II Study of Pomalidomide in Myelofibrosis With Myeloid Metaplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-4047-MMM-001
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Myelofibrosis With Myeloid Metaplasia; Myeloid Metaplasia; Myelofibrosis
Keywords: Celgene; CC-4047; Myelofibrosis; myelofibrosis with myeloid metaplasia; myeloid metaplasia; JAK2; CC-4047-MMM-001; Prednisone; Phase II; pomalidomide; bone marrow histology; imids; MMM; Ashkenazi Jewish Population; exposure to Thorotrast; exposure to solvents (benzene and toluene); acute megakaryocytic leukemia; history of polycythemia vera
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Megakaryoblastic, Acute | interventions — pomalidomide; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prednisone (Experimental): Participants received oral prednisone from Day 1-28 of each 28-day cycle for up to 3 cycles (84 days), 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day, and pomalidomide placebo tablets on Days 1-28 for up to 12 cycles in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, participants were discontinued from the study.
  Interventions: Drug: Prednisone; Drug: Placebo to pomalidomide
- Pomalidomide (Experimental): Participants received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and prednisone placebo tablets on Days 1-28 for the first 3 cycles in the Double-Blind Treatment Phase.
  After the completion of Cycle 12 and upon unblinding, participants determined to have a complete remission (CR), partial remission (PR) or clinical improvement (CI) using the International Working Group (IWG) Response Criteria in the study protocol, were eligible to participate in the extension phase and continue to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle, until disease progression, unacceptable toxicity or voluntary withdrawal.
  Interventions: Drug: Pomalidomide; Drug: Placebo to prednisone
- Pomalidomide 2 mg + Prednisone (Experimental): Participants received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, participants determined to have a complete remission (CR), partial remission (PR) or clinical improvement (CI) using the International Working Group (IWG) Response Criteria in the study protocol, were eligible to participate in the extension phase and continue to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle, until disease progression, unacceptable toxicity or voluntary withdrawal.
  Interventions: Drug: Pomalidomide; Drug: Prednisone
- Pomalidomide 0.5 mg + Prednisone (Experimental): Participants received 0.5 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, participants determined to have a complete remission (CR), partial remission (PR) or clinical improvement (CI) using the International Working Group (IWG) Response Criteria in the study protocol, were eligible to participate in the extension phase and continue to receive oral pomalidomide 0.5 mg daily, from Days 1-28 of each cycle, until disease progression, unacceptable toxicity or voluntary withdrawal.
  Interventions: Drug: Pomalidomide; Drug: Prednisone

INTERVENTIONS:
Drug: Pomalidomide
  Other Names: CC-4047; Pomalyst
  Arms: Pomalidomide; Pomalidomide 0.5 mg + Prednisone; Pomalidomide 2 mg + Prednisone
Drug: Prednisone — Participants will take oral prednisone in the evening for 3 cycles of 28 days each (up to 84 days). The dose will be as follows: 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day.
  Arms: Pomalidomide 0.5 mg + Prednisone; Pomalidomide 2 mg + Prednisone; Prednisone
Drug: Placebo to pomalidomide — Matching pomalidomide placebo tablets
  Arms: Prednisone
Drug: Placebo to prednisone — Matching prednisone placebo tablets
  Arms: Pomalidomide

SUMMARY:
The purpose of this study is to determine the safety of and to select a treatment regimen of pomalidomide (CC-4047) either as single-agent or in combination with prednisone to study further in patients with myelofibrosis with myeloid metaplasia (MMM).

DETAILED DESCRIPTION:
Participants received study treatment in the Double Blind Treatment Phase for up to 12 cycles (336 days; 12 cycles of 28 days each). Participants who completed the Double-Blind Treatment Phase were unblinded and, if receiving pomalidomide and determined to have a complete remission (CR), partial remission (PR) or clinical improvement (CI) using the International Working Group (IWG) Response Criteria in the study protocol, could have continued on their current dose of pomalidomide until disease progression. Participants receiving placebo were discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form
* Must be >18 years of age
* Must be diagnosed with myelofibrosis
* Eligibility is based on local pathology review of bone marrow aspirate and biopsy
* Screening total hemoglobin level < 10g/dL or transfusion-dependent anemia defined as per International Working Group (IWG) criteria.
* Must have adequate organ function as demonstrated by the following ≤ 14 days prior to starting study drug:

  * Alanine aminotransferase (ALT; SGPT)/aspartate aminotransferase (AST; SGOT) ≤ 3 x upper limit of normal (ULN), [unless upon judgment of the treating physician, it is believed to be due to extra-medullary hematopoiesis (EMH)].
  * Total Bilirubin <3x ULN or Direct Bilirubin <2 x ULN
  * Serum creatinine ≤ 2.0 mg/dL
  * Absolute neutrophil count ≥ 1,000/μL (≥ 1 x 10^9/L).
  * Platelet count ≥ 50,000 /μL (≥ 50 x 10^9/L).
* Patients must be willing to receive transfusion of blood products
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 at screening.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* No active malignancies with the exception of controlled prostate cancer, basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Must agree to follow pregnancy precautions as required per the protocol

Exclusion Criteria:

* Known positive status for human immunodeficiency virus (HIV), hepatitis B carrier, or active hepatitis C infection.
* Previous untoward reaction to corticosteroid (specifically, prednisone) therapy that was severe enough, in the opinion of the treating physician, to preclude study participation.
* The use of any growth factors, cytotoxic chemotherapeutic agents (e.g. hydroxyurea and anagrelide), corticosteroids, or experimental drug or therapy within a minimum of 28 days of starting CC-4047 and/or lack of recovery from all toxicity from previous therapy to grade 1 or better (e.g. alpha interferon may require 84 days of longer or washout).
* Prior therapy with CC-4047 or, lenalidomide or thalidomide for Myelofibrosis with myeloid metaplasia (MMM). (Prior prednisone use as a therapy for MMM is allowed, but not within 28 days of starting CC-4047).
* History of deep vein thrombosis or pulmonary embolism within one year of starting study medication.
* Any serious medical condition or psychiatric illness that would prevent, (as judged by the treating physician) the subject from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2009-05-01 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Peter Gale, MD, PhD, Study Director — Celgene Corporation
Locations (11):
- United States (6):
  - UCLA School of Medicine Hematology/Oncology, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian HospitalWeill Medical College of Cornell University, New York, New York
  - MD Anderson Cancer Center Leukemia Department, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Medical University of Vienna, Department of Internal Medicine, Hematology, Vienna, Austria
- Italy (2):
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - IRCCS Policlinico S. Matteo, Pavia
- Hematology DepartmentHospital Clinic, Barcelona, Spain
- Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Trust, Sheffield, United Kingdom

REFERENCES:
- [Background] Barosi G, et al. Decrease Of T Regulatory Cells In Patients With Myelofibrosis Receiving Ruxolitinib. Presented at American Society of Hematology 2013, December 7-10, 2013, New Orleans, LA. Abstract No. 4057. Blood, 2013;122(21)

RESULTS

PARTICIPANT FLOW:
Groups:
- Pomalidomide 2 mg: Participants received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and prednisone placebo tablets on Days 1-28 for the first 3 cycles in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
- Pomalidomide 2 mg + Prednisone: Participants received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
- Pomalidomide 0.5 mg + Prednisone: Participants received 0.5 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 0.5 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
Period: Overall Study
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Started | 22 | 22 | 22 | 22
Treated | 22 | 22 | 19 | 22
Completed | 0 | 0 | 0 | 0
Not Completed | 22 | 22 | 22 | 22
Not completed — Other | 4 | 3 | 6 | 4
Not completed — Adverse Event | 5 | 8 | 4 | 2
Not completed — Lack of Efficacy | 6 | 6 | 7 | 9
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Death | 2 | 1 | 2 | 0
Not completed — Missing | 2 | 0 | 0 | 2
Not completed — 1 participant received commercial drug | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone | Total
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 88
Age, Continuous [Median (Full Range); unit: years] | 66.0 [44.0 to 80.0] | 68.0 [50.0 to 83.0] | 67.5 [36.0 to 82.0] | 69.5 [43.0 to 86.0] | 67.5 [36.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 7 | 9 | 29
  Male | 14 | 17 | 15 | 13 | 59
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 22 | 21 | 22 | 86
  Black | 0 | 0 | 1 | 0 | 1
  Hispanic | 1 | 0 | 0 | 0 | 1
Janus kinase 2 (JAK2) Mutation [Number; unit: participants] — JAK2^V617F mutation result based on quantitative polymerase chain reaction (PCR) analysis in neutrophil preparation.
  participants
    Negative | 6 | 7 | 8 | 8 | 29
    Positive | 13 | 11 | 10 | 9 | 43
    Missing | 3 | 4 | 4 | 5 | 16
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance status scale and criteria used to assess disease progression, how the disease affects the daily living abilities of the patient, and determine appropriate treatment:
  0=Fully active, able to carry on all pre-disease activities;
  1. Restricted in physically strenuous activity; ambulatory and able to carry out light work;
  2. Ambulatory and capable of all selfcare; unable to perform work activities. Up and about > 50% of waking hours;
  3. Capable of only limited selfcare, confined to bed/chair > 50% of waking hours;
  4. Completely disabled. Confined to bed or chair;
  5. Dead
  participants
    Grade 0 | 12 | 11 | 6 | 14 | 43
    Grade 1 | 8 | 9 | 10 | 6 | 33
    Grade 2 | 2 | 2 | 5 | 2 | 11
    Missing | 0 | 0 | 1 | 0 | 1
Myelofibrosis with myeloid metaplasia Subtype [Number; unit: participants]
  Agnogenic Myeloid Metaplasia (AMM) | 16 | 16 | 16 | 13 | 61
  Postpolycythemic Myeloid Metaplasia (PPMM) | 3 | 4 | 4 | 2 | 13
  Postthromocythemic Myeloid Metaplasia (PTMM) | 3 | 2 | 2 | 7 | 14
Time Since Myelofibrosis Diagnosis [Median (Full Range); unit: years] | 1.5 [0.0 to 14.3] | 0.6 [0.0 to 6.3] | 1.1 [0.0 to 13.0] | 1.7 [0.0 to 10.9] | 1.1 [0.0 to 14.3]
Red Blood Cell (RBC) Transfusion Dependence [Number; unit: participants] — A patient who receives at least a total of two units of RBC transfusion within 28 days on or prior to the first study drug dosing date is an RBC-transfusion-dependent patient. Otherwise a patient is an RBC-transfusion-independent patient.
  participants
    Yes | 12 | 10 | 9 | 12 | 43
    No | 10 | 12 | 13 | 10 | 45
RBC Transfusion Burden [Median (Full Range); unit: units/28 days] | 2.0 [0.0 to 7.0] | 1.0 [0.0 to 6.0] | 0.0 [0.0 to 6.0] | 2.0 [0.0 to 4.0] | 1.0 [0.0 to 7.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinical Response Within the First 6 Cycles of Treatment
Description: A clinical responder was defined as either:
  1. A baseline red blood cell (RBC)-transfusion-dependent participant with a ≥ 56 consecutive day RBC transfusion-free period after the first dose of study drug, or
  2. A baseline RBC-transfusion-independent participant with an increase in hemoglobin of 2.0 g/dL or more from baseline for ≥ 56 consecutive days in the absence of RBC transfusions, or
  3. A participant with either a ≥ 50% reduction in palpable splenomegaly of a spleen that was ≥ 10 cm at baseline or a spleen that was palpable at > 5 cm and became not palpable.
  Participants who discontinued the study early without achieving clinical response were counted as non-responders.
Time Frame: Up to 168 days
Population: Modified intent-to-treat (MITT), defined as the patients who had a confirmed diagnosis of Myelofibrosis with myeloid metaplasia (MMM), received at least one dose of study drug, and participated in the study for at least 56 days.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 20 | 17 | 19 | 21
percentage of participants | 55.0 [31.53 to 76.94] | 23.5 [6.81 to 49.90] | 21.1 [6.05 to 45.57] | 47.6 [25.71 to 70.22]
Statistical Analysis 1: Comparison: Prednisone vs Pomalidomide 2 mg; Test type: Superiority or Other; p = 0.092, Fisher Exact
Statistical Analysis 2: Comparison: Prednisone vs Pomalidomide 2 mg + Prednisone; Test type: Superiority or Other; p = 0.048, Fisher Exact
Statistical Analysis 3: Comparison: Prednisone vs Pomalidomide 0.5 mg + Prednisone; Test type: Superiority or Other; p = 0.758, Fisher Exact

2. Secondary Outcome: Percentage of Participants With a Clinical Response Within the First 12 Cycles of Treatment
Description: as for outcome 1
Time Frame: Up to 336 days
Population: Intent-to-treat (ITT), defined as as all patients who were randomized, independent of whether they received study treatment or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 22 | 22 | 22 | 22
percentage of participants | 50.0 [28.22 to 71.78] | 18.2 [5.19 to 40.28] | 18.2 [5.19 to 40.28] | 45.5 [24.39 to 67.79]

3. Secondary Outcome: Time to the First Clinical Response
Description: The time to the first clinical response achieved within 168 days after the first study drug dosing date was calculated for participants who achieved a clinical response as:
  Start date of the first clinical response - the first study drug date +1.
  A clinical responder was defined as either:
  1. A baseline red blood cell (RBC)-transfusion-dependent participant with a ≥ 56 consecutive day RBC transfusion-free period after the first dose of study drug, or
  2. A baseline RBC-transfusion-independent participant with an increase in hemoglobin of 2.0 g/dL or more from baseline for ≥ 56 consecutive days in the absence of RBC transfusions, or
  3. A participant with either a ≥ 50% reduction in palpable splenomegaly of a spleen that was ≥ 10 cm at baseline or a spleen that was palpable at > 5 cm and became not palpable.
Time Frame: Up to 168 days
Population: Intent-to-treat population with a clinical response
Measure: Median (Full Range); unit: weeks
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 11 | 4 | 4 | 10
weeks | 0.3 [0.1 to 15.6] | 8.0 [2.6 to 17.3] | 10.1 [0.1 to 20.0] | 1.2 [0.1 to 16.6]

4. Secondary Outcome: Duration of First Clinical Response
Description: For RBC-transfusion-dependent patients, duration of response was calculated as the last day of response - first day of response +1, where the last day of response was the date of the first RBC-transfusion administrated at or more than 56 days after the response started. For patients who did not receive a subsequent transfusion after the response started, the end date of response was censored at the day of last hemoglobin assessment.
  For RBC-transfusion-independent patients, the duration of response was calculated as the last day of response - first day of response +1, where the last day of response was the earlier of the date of a hemoglobin increase of < 2.0 g/dL and the date of a RBC transfusion at ≥ 56 days after the response started. For patients whose hemoglobin measurements were always ≥ 2.0 g/dL and never received a RBC transfusion after response started, the end date of the response was censored at the date of last hemoglobin measurement.
  Kaplan-Meier methodology was used.
Time Frame: Up to 40 months
Population: Intent-to-treat population with a clinical response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 11 | 4 | 4 | 10
months | 3.7 [3.0 to 6.6] | NA [4.7 to NA] — Median not estimable as only 1 patient progressed in this group | 6.0 [2.3 to 9.8] | 10.6 [2.8 to 16.1]

5. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Anemia (FACT-An) Subscale and Total Scores
Description: The FACT-An comprises the four subscales of the 27-item FACT-General Scale (FACT-G), Physical Well-being, Social/Family Well-being, Emotion Well-being, Functional Well-Being, and the Additional Concerns Anemia subscale. Questions are rated on a scale from 0 to 4, where higher scores indicate more impact on quality of life.
  * Physical Well-being consists of 7 questions, the subscale score ranges from 0-28;
  * Social/Family Well-being consists of 7 questions, the subscale score ranges from 0-28;
  * Emotion Well-being consists of 6 questions, the subscale score ranges from 0-24;
  * Functional Well-Being consists of 7 questions, the subscale score ranges from 0-28;
  * Anemia subscale consists of 20 questions, the subscale score ranges from 0-80;
  * Total FACT-An score ranges from 0-188.
Time Frame: Baseline and Cycle 6 (168 days).
Population: Intent-to-treat patients with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 9 | 7 | 3 | 12
units on a scale
  Physical Well-Being subscale | 0.6 (1.50) | 0.4 (6.42) | 5.3 (4.04) | 2.3 (2.26)
  Social/Family Well-Being subscale | 1.9 (3.08) | -1.9 (2.59) | 1.7 (3.79) | 0.9 (6.84)
  Emotional Well-Being subscale | 1.3 (3.32) | 0.0 (4.76) | -0.3 (0.58) | 1.7 (3.47)
  Functional Well-Being subscale | 0.9 (4.14) | -2.1 (8.99) | 2.7 (3.06) | 2.5 (6.50)
  Anemia subscale | 1.2 (9.47) | 2.3 (21.34) | 19.3 (18.93) | 5.8 (8.85)
  Total FACT-An score | 2.3 (12.42) | 1.6 (36.51) | 27.3 (25.74) | 11.4 (13.51)

6. Secondary Outcome: Change From Baseline in Hemoglobin Concentration for Responders
Description: Change from Baseline in hemoglobin for participants with a clinical response within the first 6 cycles of treatment.
Time Frame: Baseline, Cycle 6 (168 days)
Population: Intent-to-treat participants with a clinical response and available hemoglobin values at each time point.
Measure: Median (Full Range); unit: g/dL
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 6 | 2 | 0 | 8
g/dL | 1.4 [-0.5 to 4.1] | 2.0 [0.7 to 3.2] |  | -0.1 [-1.9 to 3.9]

7. Secondary Outcome: Change From Baseline in Hemoglobin Concentration for Non-Responders
Description: Change from Baseline in hemoglobin for participants without a clinical response within the first 6 cycles of treatment.
Time Frame: Baseline, Cycle 6 (168 days)
Population: Intent-to-treat participants with no clinical response and available hemoglobin values at each time point.
Measure: Median (Full Range); unit: g/dL
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 3 | 5 | 5 | 6
g/dL | 1.2 [-0.2 to 2.7] | 0.1 [-0.8 to 1.3] | -0.8 [-2.0 to 1.9] | 0.5 [-0.3 to 1.0]

8. Secondary Outcome: Change From Baseline in Likert Abdominal Pain Scale
Description: Participants rated abdominal discomfort or pain over the previous week on a scale from zero to ten, where zero is no discomfort or pain and ten is the worst pain imaginable.
Time Frame: Baseline and Cycle 6 (168 days)
Population: Intent-to-treat patients with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 10 | 7 | 3 | 12
units on a scale | 0.3 (1.83) | -1.0 (3.11) | 0.3 (1.15) | -0.1 (1.68)

9. Secondary Outcome: Percentage of Participants With Clinical Response by Baseline JAK2 Assessment
Description: Percentage of participants who achieved a clinical response, presented by participants with positive and negative janus kinase 2 (JAK2) V617F mutation results at Baseline.
Time Frame: Up to 336 days
Population: Intent-to-treat population with non-missing JAK2 Baseline assessment results. The number of participants analyzed indicates the number of participants with a positive or negative JAK2 result for each treatment group respectively.
Measure: Number; unit: percentage of participants
Groups:
- Prednisone, Positive JAK2: Participants with a positive JAK2 result at Baseline received oral prednisone from Day 1-28 of each 28-day cycle for up to 3 cycles (84 days), 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day, and pomalidomide placebo tablets on Days 1-28 for up to 12 cycles in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, participants were discontinued from the study.
- Pomalidomide 2 mg, PositiveJAK2: Participants with a positive JAK2 result at Baseline received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and prednisone placebo tablets on Days 1-28 for the first 3 cycles in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
- Pomalidomide 2 mg + Prednisone, Positive JAK2: Participants with a positive JAK2 result at Baseline received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
- Pomalidomide 0.5 mg + Prednisone, Positive JAK2: Participants with a positive JAK2 result at Baseline received 0.5 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 0.5 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
- Prednisone, Negative JAK2: Participants with a negative JAK2 result at Baseline received oral prednisone from Day 1-28 of each 28-day cycle for up to 3 cycles (84 days), 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day, and pomalidomide placebo tablets on Days 1-28 for up to 12 cycles in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, participants were discontinued from the study.
- Pomalidomide 2 mg, Negative JAK2: Participants with a negative JAK2 result at Baseline received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and prednisone placebo tablets on Days 1-28 for the first 3 cycles in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
- Pomalidomide 2 mg + Prednisone, Negative JAK2: Participants with a negative JAK2 result at Baseline received 2 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 2 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
- Pomalidomide 0.5 mg + Prednisone, Negative JAK2: Participants with a negative JAK2 result at Baseline received 0.5 mg oral pomalidomide daily from Day 1-28 of each 28-day cycle for up to 12 cycles (336 days), and oral prednisone tablets on Days 1-28 for the first 3 cycles, 1st cycle = 30 mg daily, 2nd cycle = 15 mg daily, 3rd cycle = 15 mg every other day in the Double-Blind Treatment Phase.
  After the completion of cycle 12 and upon unblinding, eligible participants continued to receive oral pomalidomide 0.5 mg daily, from Days 1-28 of each cycle. Participants could remain on study treatment in the Extension Phase until disease progression, unacceptable toxicity or voluntary withdrawal.
Arm/Group | Prednisone, Positive JAK2 | Pomalidomide 2 mg, PositiveJAK2 | Pomalidomide 2 mg + Prednisone, Positive JAK2 | Pomalidomide 0.5 mg + Prednisone, Positive JAK2 | Prednisone, Negative JAK2 | Pomalidomide 2 mg, Negative JAK2 | Pomalidomide 2 mg + Prednisone, Negative JAK2 | Pomalidomide 0.5 mg + Prednisone, Negative JAK2
Number analyzed (Participants) | 13 | 11 | 10 | 9 | 6 | 7 | 8 | 8
percentage of participants | 46.2 | 27.3 | 30.0 | 66.7 | 50.0 | 28.6 | 12.5 | 25.0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious AE (SAE) was defined as any AE which resulted in death or was life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or constituted an important medical event (events that may have jeopardized the patient or required intervention to prevent one of the outcomes listed above).
  The severity of AEs were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 3.0) or according to the following scale:
  Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening; Grade 5 = Death.
  The Investigator determined the relationship between study drug and the occurrence of an AE as "Not Related" or "Related" (since the study was double-blinded, a patient receiving only prednisone could have an AE that was judged as related to pomalidomide, and vice-versa).
Time Frame: From date of the first dose of the study drug until discontinuation or the data cut-off date (up to approximately 45 months).
Population: Safety population (all treated patients).
Measure: Number; unit: participants
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Number analyzed (Participants) | 22 | 22 | 19 | 22
participants
  At least one AE | 20 | 21 | 18 | 21
  At least one AE related to pomalidomide | 15 | 17 | 16 | 15
  At least one AE related to prednisone | 10 | 10 | 11 | 5
  At least one Grade 3-4 AE | 10 | 14 | 13 | 15
  At least one Grade 3-4 AE related to pomalidomide | 6 | 7 | 11 | 6
  At least one Grade 3-4 AE related to prednisone | 5 | 2 | 6 | 3
  At least one SAE | 6 | 10 | 11 | 8
  At least one SAE related to pomalidomide | 4 | 6 | 8 | 3
  At least one SAE related to prednisone | 4 | 3 | 5 | 3
  AE leading to discontinuation of pomalidomide | 7 | 11 | 5 | 6
  AE leading to discontinuation of prednisone | 5 | 7 | 2 | 1
  AE leading to a dose reduction of pomalidomide | 0 | 2 | 1 | 1
  AE leading to a dose interruption of pomalidomide | 5 | 9 | 9 | 7
  AE leading to a dose interruption of prednisone | 2 | 8 | 6 | 3

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug through to 30 days after the last dose; up to the data cut-off date of 18 December 2013; up to 81 months
Arm/Group | Prednisone | Pomalidomide 2 mg | Pomalidomide 2 mg + Prednisone | Pomalidomide 0.5 mg + Prednisone
Serious Adverse Events (participants affected / at risk) | 6/22 | 10/22 | 11/19 | 9/22
Other Adverse Events (participants affected / at risk) | 20/22 | 20/22 | 17/19 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone (N=22) | Pomalidomide 2 mg (N=22) | Pomalidomide 2 mg + Prednisone (N=19) | Pomalidomide 0.5 mg + Prednisone (N=22)
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 3 | 2
Septic Shock (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Lung Infection Pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Perirectal Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Varices Oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Disease Progression (General disorders) | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 2 | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Acquired Von Willebrand Disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone (N=22) | Pomalidomide 2 mg (N=22) | Pomalidomide 2 mg + Prednisone (N=19) | Pomalidomide 0.5 mg + Prednisone (N=22)
Fatigue (General disorders) | 6 | 2 | 6 | 7
Oedema Peripheral (General disorders) | 6 | 8 | 10 | 10
Pyrexia (General disorders) | 5 | 7 | 4 | 6
Chills (General disorders) | 2 | 2 | 1 | 4
Asthenia (General disorders) | 1 | 3 | 1 | 4
Feeling Jittery (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 4 | 8
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5 | 3
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 7 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 3 | 1 | 5
Nausea (Gastrointestinal disorders) | 4 | 4 | 3 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 2 | 5 | 4
Oral Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 1 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 5 | 3
Gingival Bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Tongue Ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 2 | 6 | 8
Paraesthesia (Nervous system disorders) | 4 | 2 | 3 | 4
Burning Sensation (Nervous system disorders) | 3 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 2 | 0 | 4
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 2
Memory Impairment (Nervous system disorders) | 1 | 1 | 2 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2 | 1 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 2 | 2
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1
Enterococcal Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 3
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Increased Tendency To Bruise (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 8 | 3 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 4
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Odour Abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 2 | 2 | 3
Depression (Psychiatric disorders) | 1 | 2 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 2 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 1 | 0
Personality Change (Psychiatric disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 3 | 2 | 4 | 1
Eye Irritation (Eye disorders) | 0 | 1 | 2 | 1
Lacrimation Increased (Eye disorders) | 0 | 0 | 2 | 0
Periorbital Oedema (Eye disorders) | 0 | 0 | 1 | 1
Heart Rate Increased (Investigations) | 2 | 0 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 0 | 2
Cardiac Murmur (Investigations) | 0 | 2 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 1
Ear Congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 2 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 3 | 0 | 0
Gait Disturbance (General disorders) | 0 | 2 | 0 | 0
Oedema (General disorders) | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally thirty (60) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.